CLINICAL TRIAL: NCT06029803
Title: Antecubital Versus Femoral Approach for Adrenal Venous Sampling: A Randomised Controlled Trial
Brief Title: Antecubital Versus Femoral Approach for Adrenal Venous Sampling
Acronym: AFAVS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Principal Investigator, Hui DONG, professor, Chinese Academy of Medical Sciences, Fuwai Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2022-1715
Record Dates: First submitted 2023-08-26; First posted 2023-09-08 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-09

CONDITIONS: Hyperaldosteronism
Keywords: Adrenal venous sampling; Hyperaldosteronism; Antecubital approach; Femoral approach
MeSH Terms: conditions — Hyperaldosteronism

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adrenal Venous Sampling via Antecubital Approach (Experimental): Patients in the experimental group will undergo adrenal venous sampling via antecubital vein approach.
  Interventions: Procedure: Adrenal Venous Sampling via Antecubital Approach
- Adrenal Venous Sampling via Femoral Approach (Active Comparator): Patients in the active comparator group will undergo adrenal venous sampling via femoral vein approach.
  Interventions: Procedure: Adrenal Venous Sampling via Femoral Approach

INTERVENTIONS:
Procedure: Adrenal Venous Sampling via Antecubital Approach — Patients assigned to the antecubital approach group (experimental group) will undergo AVS via antecubital approach.A 5F introducer sheath will be introduced into the antecubital vein. After heparinization,a diagnostic catheter with side holes will be introduced. Two blood samples (about 4mL each) will be collected from the inferior vena cava, right adrenal vein and left adrenal vein for the determination of cortisol and aldosterone concentrations.
  Arms: Adrenal Venous Sampling via Antecubital Approach
Procedure: Adrenal Venous Sampling via Femoral Approach — Patients assigned to the femoral approach group (active comparator group) will undergo AVS via femoral vein approach.The introducer sheath will be introduced into the femoral vein.Two blood samples (about 4mL each) will be collected from the inferior vena cava, right adrenal vein and left adrenal vein for the determination of cortisol and aldosterone concentrations.
  Arms: Adrenal Venous Sampling via Femoral Approach

SUMMARY:
Subtype diagnosis is crucial for the treatment of primary aldosteronism (PA), which conducts the appropriate treatment strategy. Currently, adrenal venous sampling (AVS) serves as the gold standard for subtyping of PA. At present, almost all medical centers use the femoral vein approach for AVS, and most studies report that the success rate is 30%-80%. Our research team is the first in the world to conduct AVS via an antecubital approach. The aim of this study is to compare the success rate and safety of AVS via antecubital and femoral approach.

DETAILED DESCRIPTION:
Primary aldosteronism (PA) is one of the most common causes of secondary hypertension, and its most common subtypes are aldosterone-producing adenoma and idiopathic hyperaldosteronism, which account for 95% to 98% of PA. Subtype diagnosis is crucial for the treatment of primary aldosteronism, which conducts the appropriate treatment strategy. Currently, adrenal venous sampling (AVS) serves as the gold standard for subtyping of PA. At present, almost all medical centers use the femoral vein approach for AVS, and most studies report that the success rate is 30%-80%.How to improve the success rate of AVS has been a hot topic in the field of primary aldosteronism. Our research team is the first in the world to conduct AVS via an antecubital approach. The previous study found that the success rate of AVS via this approach can reach to 88.0%, with a low incidence of complications. In this study, patients with primary aldosteronism who meet the indications of AVS will be randomly assigned to antecubital approach group and femoral approach group. Clinical, laboratory and examination data will be recorded and the success rate and safety of AVS via antecubital and femoral approach will be compared.

ELIGIBILITY:
Inclusion Criteria:

1. Aged from 18 to 60 with no limits in sex;
2. Patients with confirmed primary aldosteronism;
3. Patients or their legal representatives sign written informed consent approved by the ethics committee

Exclusion Criteria:

1. Severe comorbidity, including stroke, myocardial infarction, heart failure, severe valvular heart disease, liver cirrhosis, and metastatic tumor within the previous 3 months；
2. An estimated glomerular filtration rate <45 ml/min/1.73 m2, or serum creatinine >176 μmol/L；
3. Patients who refuse adrenalectomy;
4. suspected of having an adrenocortical carcinoma;
5. allergy to contrast agent;
6. pregnant, nursing, or planning to become pregnant

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 154 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-11-30 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
The success rate of bilateral adrenal venous sampling | At AVS procedure
  Successful sampling will be defined by high selectivity index (cortisol in the adrenal vein/cortisol in inferior vena cava >2 without ACTH simulation)

SECONDARY OUTCOMES:
The success rate of left adrenal venous sampling | At AVS procedure
  Successful sampling will be defined by high selectivity index (cortisol in the adrenal vein/cortisol in inferior vena cava >2 without ACTH simulation)
The success rate of right adrenal venous sampling | At AVS procedure
  Successful sampling will be defined by high selectivity index (cortisol in the adrenal vein/cortisol in inferior vena cava >2 without ACTH simulation)
Selection of intraoperative catheter | At AVS procedure
  Catheter selection
Time of the procedure | At AVS procedure
  Time of the procedure
Time of fluoroscopy | At AVS procedure
  Time of fluoroscopy
The contrast agent dosage | At AVS procedure
  The contrast agent dosage
the incidence of complications | 1 week after AVS procedure
  Complications related to adrenal vein cannulations (adrenal vein hematoma, inferior vena cava dissection, puncture site hematoma, etc)
the cost of the procedure | At AVS procedure
  the cost of the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Hui Dong, MD, Principal Investigator — Fuwai Hospital, National Center for Cardiovascular Disease, Chinese Academy of Medical Sciences and Peking Union Medical College
Locations (1):
- Fuwai Hospital, National Center for Cardiovascular Disease, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, Beijing Municipality, China